CLINICAL TRIAL: NCT05892003
Title: Healthy Diets for a Healthy Weight: Exploring Physiological Mechanisms Related to Dietary Fibre and Non-Nutritive Sweeteners
Brief Title: Scot Sweet Study (Interaction of a Non-nutritive Sweetener With a High-fibre Weight Loss Diet)
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 814
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Appetitive Behavior
Keywords: fibre; non-nutritive sweetener; weight loss; gut microbiome; glycaemic control
MeSH Terms: conditions — Appetitive Behavior; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control-High Fibre Weight Loss-High Fibre Non-Nutritive Sweetener Weight Loss: CTRL-HF WL-HF-NNS WL (Experimental): * Phase 1 CTRL: Control diet with moderate fibre consumption for 14days.
  * Phase 2 HF WL: High Fibre Weight Loss meal consumption for 14days.
  * Phase 3 HF-NNS WL: High Fibre and Non-Nutritive Sweetener Weight Loss meal consumption for 14days.
  Interventions: Other: Phase 1 Control; Other: Phase 2 High Fibre Weight Loss; Other: Phase 3 High Fibre and Non-Nutritive Sweetener Weight Loss

INTERVENTIONS:
Other: Phase 1 Control — Control diet (30% Fat, 15% Protein, 55% Carbohydrate, Fibre rising from 10 to 16g/d). Fed to energy balance (1.5 x Resting Metabolic Rate, RMR).
  Other Names: CTRL
Other: Phase 2 High Fibre Weight Loss — High Fibre Weight Loss diet (30% Fat, 15% Protein, 55% Carbohydrate). Fed to energy deficit (100% RMR). The quantity of fructo-oligosaccharides (FOS) will be fixed at 20g/day for all kcal levels with additional fibre coming from the diet provided. The FOS will be split over breakfast, lunch and dinner in drinks/yoghurts which will be compulsory to consume.
  Other Names: HF WL
Other: Phase 3 High Fibre and Non-Nutritive Sweetener Weight Loss — High Fibre and Non-Nutritive Sweetener Weight Loss diet (30% Fat, 15% Protein, 55% Carbohydrate). Fed to energy deficit (100% RMR). The quantity of fructo-oligosaccharides (FOS) and non-nutritive sweetener (sucralose) will be fixed at 20g/day and 30mg/day respectively for all kcal levels with additional fibre coming from the diet provided. The FOS and sucralose will be split over breakfast, lunch and dinner in drinks/yoghurts which will be compulsory to consume.
  Other Names: HF-NNS WL

SUMMARY:
The investigators present a weight loss diet intervention study, to be conducted as a within-subject design, with all food and beverages provided, to assess interaction of non-nutritive sweetener (sucralose) with a high-fibre weight loss diet, on markers of gut health in humans. This study will allow assessment of the effects of a non-nutritive sweetener (sucralose) with a high-fibre (soluble fibre, fructo-oligosaccharides, FOS) diet on metabolic health and activity and composition of gut microbiota, by a controlled human diet intervention study. The investigators propose to recruit participants living with obesity, with a poor diet quality (moderate habitual fibre intake) to additionally address diet inequalities in the research approach, and this will also allow examine the time-course of adaptation of the gut microbiome (measured in faecal samples). The investigators will also assess changes in free-living glycaemic control with addition of dietary fibre and bio-markers of health.

ELIGIBILITY:
Inclusion Criteria:

* healthy but overweight/obese (BMI 28-40kg/m2) males and females (postmenopausal, using the oral contraceptive pill or some form of hormonal contraceptive)
* moderate habitual fibre intake (18-23g/day)

Exclusion Criteria:

Medication exclusion criteria:

* antibiotic use (within the past 3 months due to impact on gut microbiota)
* anti-depressants (current)
* smoking or vaping
* weight loss medication

Medical exclusion criteria:

* Females who are planning to be pregnant, are pregnant or are breastfeeding
* Anyone with food allergies, self-reported food sensitivity or intolerance
* Anyone with coeliac disease or gluten intolerance
* Anyone taking medication which may affect their appetite
* Anyone with an eating disorder
* Anyone with diabetes
* Anyone with a gastrointestinal disorder, kidney disease, liver disease or gout
* Anyone suffering from a psychiatric disorder or any type of substance abuse
* Anyone suffering from unregulated thyroid disease

Other exclusion criteria:

* Anyone following a vegetarian or vegan diet
* Anyone following a current weight loss programme (that may be affecting lifestyle, physical activity & diet) or undergone gastric band/reduction surgery
* Anyone with unsuitable veins for blood sampling
* Anyone who is unable to fluently speak, read and understand English
* Anyone who is unable to comply to an alcohol-free diet for 6 weeks

Current sweetener consumption will not be an exclusion criteria as the Phase 1 - CTRL and Phase 2 - HF WL diets will provide enough of a washout (4 weeks) before the Phase 3 diets containing sucralose are consumed. Participants who do habitually consume sweeteners will be asked not to use them during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in gut metabolites (from faecal samples) in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  Measured by changes in faecal short chain fatty acids concentrations
Change in gut microbiome composition (from faecal samples) in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  Measured by changes in bacterial 16S ribosomal ribonucleic acid gene sequencing; 16S rRNA
Change in gut metabolite production (from faecal samples) in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  Measured by changes in calprotectin concentrations

SECONDARY OUTCOMES:
Change in free-living glycaemic control in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured using continuous glucose monitoring (CGM)
Change in glycaemic control in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  measured by changes in fasted plasma glucose and insulin

OTHER OUTCOMES:
Change in concentration of blood metabolites in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  measured by changes in fasted plasma short chain fatty acid (SCFA) concentrations
Change in concentration of gut hormones in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  measured by changes in fasted plasma ghrelin, GLP-1 and peptide YY (PYY) concentrations
Change in lipid profile in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  measured by changes in fasted plasma lipid profile (Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and non-esterified fatty acids (NEFA)
Change in lipid ratios in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  Total cholesterol, HDL-cholesterol and LDL-cholesterol measures will be combined to report TC to HDL and LDL to HDL ratios.
Change in concentration of urinary metabolites in response to dietary fibre and non-nutritive sweetener | At baseline and end of each arm (study days 1, 15, 29 and 43)
  changes in urinary metabolite concentrations measured by metabolomics
Height | At screening visit only
  measured in metres
Change in body weight in response to dietary fibre and non-nutritive sweetener | At screening and 3 times a week on each arm (20 occasions from date of screening up to study day 43)
  measured as weight in kilograms
Change in Body Mass Index (BMI) in response to dietary fibre and non-nutritive sweetener | At screening and 3 times a week on each arm (20 occasions from date of screening up to study day 43)
  weight and height measures will be combined to report BMI in kg/m^2
Change in daily nausea symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced nausea today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily bloating symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced bloating today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily flatulence symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced flatulence today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily abdominal cramp symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced abdominal cramps today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily intestinal rumble symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced rumbles today? (intestinal sounds)', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily diarrhoea symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced diarrhoea today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily constipation symptoms in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a Likert scale 'Have you experienced constipation today?', scored as 0 - no more symptoms than usual, 1 - slightly more symptoms than usual, 2 - noticeably more symptoms than usual, 3 - considerably more symptoms than usual.
Change in daily bowel movements in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a scale 'How many bowel movements have you had today?', scored as 0, 1, 2, 3 or >3.
Change in daily hunger rating in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a visual analogue scale 'How hungry have you felt today?', scored from 0 (Generally not at all hungry) to 100 (Generally as hungry as I've ever felt).
Change in daily fullness rating in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a visual analogue scale 'How full have you felt today?', scored from 0 (Generally not at all full) to 100 (Generally as full as I've ever felt).
Change in daily desire to eat rating in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a visual analogue scale 'How strong has your desire to eat been today?', scored from 0 (Very weak) to 100 (Very strong).
Change in retrospective food consumption rating in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  measured daily, at end of day, using questionnaires. Question presented as a visual analogue scale 'How much do you feel you could have eaten today?', scored from 0 (Nothing at all) to 100 (A large amount).
Change in appetite in response to dietary fibre and non-nutritive sweetener | every day of study diets (42days)
  Mean of hunger, fullness, desire to eat and retrospective consumption ratings will be combined to report an overall appetite score (from 0 to 100)
Change in food intake | at screening (7days) and every day of study diets (42days)
  measured using weighed intake records

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, Prof, Principal Investigator — Rowett Institute, University of Aberdeen; Alexander Ross, Dr, Principal Investigator — Rowett Institute, University of Aberdeen
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No